CLINICAL TRIAL: NCT04146064
Title: Breathomics as a Non-invasive, Inexpensive, Point-of-care Predictive Test for Immune Checkpoint Inhibitor Efficacy
Brief Title: Breathomics as Predictive Biomarker for Checkpoint Inhibitor Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Amsterdam (Other)
Responsible Party: Sponsor
Other Study IDs: IO-Breathomics; 19-5936 (Other: CAPCR-University Health Network)
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: NSCLC; Melanoma; Kidney Cancer; Urothelial Carcinoma; Head and Neck Cancer
Keywords: breathprint analysis; immunotherapy; predictive biomarker
MeSH Terms: conditions — Melanoma; Kidney Neoplasms; Carcinoma, Transitional Cell; Head and Neck Neoplasms | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Validation cohort: NSCLC: Patients with advanced/metastatic NSCLC planned for IO-treatment in one of the following categories
  * Pembrolizumab monotherapy first-line
  * Pembrolizumab or nivolumab monotherapy in second or later line
  Interventions: Other: Breathprint analysis and patient-reported outcomes
- Cohort 1: NSCLC: Patients with advanced/metastatic NSCLC planned for Pembrolizumab-chemotherapy combination therapy first-line
  Interventions: Other: Breathprint analysis and patient-reported outcomes
- Cohort 2: Melanoma: Patients with advanced/metastatic melanoma planned for IO-treatment in one of the following categories
  * Nivolumab/ipilimumab combination treatment 1L
  * Pembrolizumab or nivolumab monotherapy treatment 1L
  * Ipilimumab monotherapy 2L
  Interventions: Other: Breathprint analysis and patient-reported outcomes
- Cohort 3: Mixed solid tumor cohort: Patients with advanced/metastatic solid tumors such as Head&Neck tumors, kidney cancer and urothelial cancer planned for IO-treatment
  Interventions: Other: Breathprint analysis and patient-reported outcomes
- Cohort 4: NSCLC: Patients with advanced/metastatic NSCLC planned for treatment with Chemotherapy-only (either platinum-based combination treatment or docetaxel monotherapy)
  Interventions: Other: Breathprint analysis and patient-reported outcomes

INTERVENTIONS:
Other: Breathprint analysis and patient-reported outcomes — Breathprint analysis: Patients will be providing breathprint samples into the eNose device at baseline and every 12 weeks thereafter as long as on immunotherapy treatment.
  Questionnaires will be completed at the same timepoints.

SUMMARY:
Immunotherapy with agents stimulating the immune system to act against cancer are now a new standard of care in various cancers as lung cancer and melanoma, but also bladder cancer, kidney cancer and head & neck cancer. However, even though a subset of patients derives long-term benefit from these agents, depending of cancer type still at least half of patients do not respond to these new drugs. Our understanding of possible factors predicting whether a patient might actually benefit from immunotherapy is poor. Volatile organic compounds (VOCs) are gases exhaled with a person's breath, which are released into the lung from blood and bacteria and therefore can give information about infections as well as inflammation and possibly cancer cells in a person's body. Breath analysis of these VOCs with special devices called electronic noses (eNose) generate a specific electric signals patterns called breathprints. There is early evidence that specific breathprints can actually help to select patients who will be likely to benefit from immunotherapy.

This study is being undertaken in an effort to evaluate breathprint analysis as a potential predicting factor for benefit from immunotherapy, so that treatment selection can further be improved.

This study is designed to help us identify the role of breathprint analysis to better select patients for immunotherapy.

DETAILED DESCRIPTION:
Immune checkpoint blockade with anti-PD-1 and anti-PD-L1 antibodies has become a new standard of care in several cancer types as NSCLC and melanoma. However, in biomarker-unselected patient populations, overall response rate (ORR) depending on type of cancer and whether single or combination treatment is chosen remains still only 20%-60%. Though overall well tolerated approximately 5-10% of patients treated with PD1/PD-L1 targeting agents will experience grade 3 or 4 toxicities, including potentially life-threatening auto-immune toxicities such as colitis, hepatitis, and pneumonitis. Therefore, due to high costs of treatment and its possible complications, improved selection of patients is a crucial goal and an easily available non-invasive, point-of-care test for better patient selection is very much needed.

A promising approach in this regard is the analysis of volatile organic compounds (VOCs) in breath. Breath analysis for the detection of VOCs is increasingly investigated for its utility in diagnosis and management of cancer. Electronic noses (eNoses) are promising as cheap and clinically-practical devices that are designed to detect patterns of VOCs. Recently published prospective observational data showed very promising discriminant function for breathprint analysis for non-response to immunotherapy in NSCLC patients.

The principle goal of this study is to validate a prior study that found that breathomics-based classifiers predicted 12-week early progression vs non-progression in advanced NSCLC patients treated with nivolumab or pembrolizumab. Secondarily, we will expand assessment of breathomic-based classifiers to include other cohorts of advanced tumors treated with ICI, and also consider using response instead of non-progression as an endpoint. Exploratory goals include refinement of the breathomics classifier using alternative machine-learning techniques, and correlate with other biomarkers of immunotherapy outcomes.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients 18 years of age or older
* Histologically confirmed advanced/metastatic non-small cell lung cancer, melanoma or solid tumor such as urothelial, kidney or head and neck cancer and planned treatment with

  * NSCLC validation cohort: Pembrolizumab or Nivolumab
  * NSCLC Cohort 1: Pembrolizumab-chemotherapy combination therapy 1L
  * Melanoma Cohort 2: Nivolumab/ipilimumab combination treatment 1L, Pembrolizumab or nivolumab monotherapy treatment 1L , Ipilimumab
  * Solid tumors Cohort 3: Any ICI-treatment, any line
  * NSCLC Cohort 4: Chemotherapy-only (either platinum-based combination treatment or docetaxel monotherapy)
* At least one measurable lesion as defined by RECIST 1.1. A lesion at a previously irradiated site may only be counted as a target lesion if there is clear sign of progression since the irradiation.
* Able to provide informed consent.

EXCLUSION CRITERIA

* Patients who are unable to perform the breathing manoeuvres needed for eNose-analysis of exhaled air.
* Patients who are unable to independently consent to participation in the trial.
* Patients with severe, acute, or chronic medical conditions (including uncontrolled diabetes mellitus) or psychiatric conditions or laboratory abnormalities that in the opinion of the Investigator or their physician may cause undue harm or inconvenience to the patient, or that may interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in this study are patients over the age of 18 years with a histologically-confirmed diagnosis of non-small cell lung cancer, melanoma or other solid tumor for which ICI-treatment is a standard of care. Patients must have advanced/metastatic disease and planning to receive ICI treatment (categories defined above) or chemotherapy treatment (cohort 4) at the Princess Margaret Cancer Centre/University Health Network. Study subjects will be consented specifically for that study.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
12 week Progression Rate in validation cohort | 12 weeks

SECONDARY OUTCOMES:
Overall Survival (OS) in validation cohort | 5 years
Overall Response Rate (ORR) in validation cohort | 5 years

OTHER OUTCOMES:
Progression-free survival (PFS) in validation cohort | 5 years
6 months clinical benefit rate (CR, PR or SD at 6 months after treatment start) in validation cohort | 6 months
12 week Progression Rate in exploratory cohorts | 12 weeks
OS in exploratory cohorts | 5 years
Overall Response Rate (ORR) in exploratory cohorts | 5 years
PFS in exploratory cohorts | 5 years
6 months clinical benefit rate in exploratory cohorts | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Liu, MD MSc, Principal Investigator — UHN
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided